CLINICAL TRIAL: NCT00768664
Title: CLINICAL PHASE 2 MULTICENTER TRIAL OF PF-00299804 IN PATIENTS WITH RECURRENT OR METASTATIC SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK
Brief Title: Open-Label Trial Of Oral PF-00299804 By Continuous Dosing In Patients With Recurrent Or Metastatic Head And Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471027
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Head and Neck Neoplasms
Keywords: recurrent or metastatic squamous cell cancer of the Head and Neck; no prior systemic therapy for recurrence
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — 45 mg by continuous oral dosing

SUMMARY:
This study will investigate the safety and efficacy of oral PF-00299804 in patients who have not yet undergone any other drug treatment for recurrent and/ or metastatic head and neck squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic Squamous Cell Cancer of the Head and Neck;
* Measurable disease;
* Eastern Cooperative Oncology Group (ECOG) 0-1 in Stage 1 = first 23 patients;
* Eastern Cooperative Oncology Group (ECOG) 0-2 in Stage 2 = 33 patients;

Exclusion Criteria:

* prior therapy for recurrence;
* platelets < 75,000;
* prior Epidermal Growth Factor Receptor (EGFR) therapy;
* interstitial lung disease;
* primary of nasopharynx

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-11-04 (Actual); Primary Completion 2010-05-05 (Actual); Study Completion 2012-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Canada (9):
  - BC Cancer Agency, Vancouver Centre, Vancouver, British Columbia
  - Fairmont Medical Building, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - London Regional Cancer Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre: Odette Cancer Center, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-dame du CHUM - Oncology Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471027&StudyName=Open-Label%20Trial%20Of%20Oral%20PF-00299804%20By%20Continuous%20Dosing%20In%20Patients%20With%20Recurrent%20Or%20Metastatic%20Head%20And%20Neck%20Squamous%20Cell%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Dacomitinib 45 mg: Participants with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) received dacomitinib 45 milligram (mg) tablets, orally, once daily (QD) continuously until unacceptable toxicity, disease progression, withdrawal of consent, or death. There were no planned treatment breaks, each cycle was defined as 21 days for the purposes of scheduling. Dose reductions (in 15 mg increments) to a minimum of 15 mg QD were allowed; dose re-escalations were not allowed.
Period: Overall Study
Arm/Group | Dacomitinib 45 mg
Started | 69
Completed | 0
Not Completed | 69
Not completed — Death | 57
Not completed — Lost to Follow-up | 2
Not completed — Other | 9
Not completed — Participant refused | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR) of Complete Response (CR) or Partial Response (PR)
Description: Percentage of participants with best OR of confirmed CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) relative to total number of evaluable participants for response. CR defined as disappearance of all target/non-target lesions. PR defined as at least a 30 percent (%) decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions. Confirmed responses (CR and PR) were those that persisted on a follow-up imaging assessment greater than or equal to (≥)4 weeks after the initial objective documentation of response.
Time Frame: Baseline up to 18 months
Population: Response-Evaluable Population: All participants with measurable disease (per RECIST), treated, with baseline and ≥1 on-study assessment. Participants who discontinued early before on-study tumor assessment due to PD were evaluable, but not if discontinued early due to reasons such as participant request, lack of compliance, or early toxicity.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 63
Percentage of participants | 12.5 [5.6 to 23.5]

2. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response (CR or PR) to progression or death due to progressive disease (PD). DR was calculated as (the date of the first documentation of PD or death due to PD minus the date of the first CR or PR that was subsequently confirmed plus 1). DR was calculated for the subgroup of participants with a confirmed objective tumor response (CR or PR).
Time Frame: Baseline up to 18 months
Population: Response Evaluable population; n equals (=) number of participants with an objective response of CR or PR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 8
weeks | 17.9 [12.6 to 20.1]

3. Secondary Outcome: Duration of Stable Disease (SD)
Description: Time in weeks from start of treatment to date of objective disease progression (based on RECIST criteria). SD defined as neither sufficient shrinkage for PR nor sufficient increase for PD, taking as a reference the smallest sum of the longest dimensions since treatment start. Participants last known to be alive, not to have started new anticancer treatment, to be progression free, and who had a baseline and at least 1 on-study disease assessment were censored at date of last objective disease assessment that verified lack of PD. Participants who died not due to PD censored on death date.
Time Frame: Baseline up to 18 months
Population: Response Evaluable population; n=number of participants with a best overall response of SD.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 36
weeks | 14.6 [12.0 to 24.7]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in weeks from date of enrollment to first documentation of PD, death due to any cause, symptomatic deterioration, or start of secondary anticancer therapy, whichever occurred first. PFS calculated as (first event date minus enrollment date plus 1). Documentation of progression determined from objective disease assessment based on RECIST criteria. PD defined as at least a 20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since treatment started or the appearance of 1 or more new lesions.
Time Frame: Baseline up to 18 months
Population: ITT Population: all enrolled participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 69
weeks | 12.1 [11.1 to 17.9]

5. Secondary Outcome: Progression-Free Survival (PFS) at 6 Months and at 1 Year
Description: Probability of being event-free (event defined as PD, death due to any cause, symptomatic deterioration, or start of secondary anticancer therapy) at 26 weeks and 52 weeks after the first dose of study treatment.
Time Frame: Baseline up to 52 weeks
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percent chance of being event free
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 69
percent chance of being event free
  Probability of being event free at Week 26 | 21.4 [11.4 to 33.4]
  Probability of being event free at Week 52 | 2.1 [0.2 to 9.8]

6. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from the start date of enrollment to date of death due to any cause. OS was calculated as (the death date minus the enrollment date plus 1). Participants without death dates, last known to be alive were censored at last contact.
Time Frame: Baseline up to 18 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 69
weeks | 34.6 [29.4 to 52.1]

7. Secondary Outcome: Overall Survival at 6 Months and 1 Year
Description: Probability of survival 26 weeks and 52 weeks after the first dose of study treatment.
Time Frame: Baseline up to Week 52
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percent chance of survival
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 69
percent chance of survival
  Survival Probability at Week 26 | 66.5 [53.7 to 76.5]
  Survival Probability at Week 52 | 39.6 [27.6 to 51.3]

8. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of Dacomitinib After Repeat Dosing
Description: Trough concentrations of dacomitinib in plasma measured as nanograms per milliliter (ng/mL).
Time Frame: Predose on Day 1 of Cycles 2, 3, and 4 and predose on Day 8 of Cycle 1
Population: Pharmacokinetic (PK) population: all enrolled participants who received at least 1 dose of study medication from whom at least 1 PK sample was obtained. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for specific rows.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 63
ng/mL
  Cycle 1 Day 8 | 64.30 [0.000 to 118]
  Cycle 2 Day 1: number analyzed (Participants) | 60
  Cycle 2 Day 1 | 76.85 [7.67 to 244]
  Cycle 3 Day 1: number analyzed (Participants) | 43
  Cycle 3 Day 1 | 74.50 [21.6 to 248]
  Cycle 4 Day 1: number analyzed (Participants) | 39
  Cycle 4 Day 1 | 69.60 [12.1 to 191]

9. Secondary Outcome: Ctrough of Dacomitinib After Repeat Dosing In Participants Requiring Administration of Dacomitinib With a Feeding Tube
Time Frame: Predose on Day 1 of Cycles 2, 3, and 4 and predose on Day 8 of Cycle 1
Population: PK population: all enrolled participants who received at least 1 dose of study medication from whom at least 1 PK sample was obtained. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for specific rows.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Day 8 | 81.30 [46.1 to 105]
  Cycle 2 Day 1: number analyzed (Participants) | 6
  Cycle 2 Day 1 | 92.05 [64.3 to 130]
  Cycle 3 Day 1: number analyzed (Participants) | 2
  Cycle 3 Day 1 | 129.2 [95.3 to 163]
  Cycle 4 Day 1: number analyzed (Participants) | 1
  Cycle 4 Day 1 | 156 [156 to 156]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) In Participants Requiring Administration of Dacomitinib With a Feeding Tube
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, 6, 8, 10, and 24 hours postdose
Population: PK Population; n=number of participants requiring administration of dacomitinib with a feeding tube.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 1
ng/mL | 23.80 [23.8 to 23.8]

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) In Participants Requiring Administration of Dacomitinib With a Feeding Tube
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, 6, 8, 10, and 24 hours postdose
Population: PK Population; n=number of participants requiring administration of dacomitinib with a feeding tube.
Measure: Median (Full Range); unit: ng*hour (hr)/mL
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 1
ng*hour (hr)/mL | 285.0 [285 to 285]

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) In Participants Requiring Administration of Dacomitinib With a Feeding Tube
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, 6, 8, 10, and 24 hours postdose
Population: PK Population; n=number of participants requiring administration of dacomitinib with a feeding tube.
Measure: Median (Full Range); unit: hours
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 1
hours | 4.00 [4.00 to 4.00]

13. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Cycle 1 Day 1 at predose and 1, 2, 4, 6, 8, 10, and 24 hours postdose
Population: PK Population; n=number of participants requiring administration of dacomitinib with a feeding tube.
Measure: Median (Full Range); unit: hours
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 1
hours | NA [NA to NA] — Insufficient sampling to determine plasma half-life

14. Secondary Outcome: Correlation Between Biomarkers Status and Best Overall Response
Description: The best overall response was best response recorded from the start of the treatment until disease progression/recurrence. In this outcome measure, biomarkers status and best overall response was reported in terms of correlation coefficient.
Time Frame: Baseline up to 18 months
Population: Biomarker analysis set: all enrolled participants who had baseline samples submitted as per Institutional Review Board/Independent Ethics Committee approval and participant consent. Here, "number analyzed" signifies participants evaluable at specific rows.
Measure: Number; unit: Correlation coefficient
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 48
Correlation coefficient
  HPV Overall Status: number analyzed (Participants) | 41
  HPV Overall Status | 0.799
  EGFR VIII Status with DNA Method: number analyzed (Participants) | 40
  EGFR VIII Status with DNA Method | 1.000
  PTEN:: number analyzed (Participants) | 38
  PTEN: | 0.840
  Mutation: number analyzed (Participants) | 44
  Mutation | 1.000

15. Secondary Outcome: H-Score at Baseline and Post-baseline for Paired Biopsy Biomarkers
Description: H-score is a measure of the immunohistochemistry staining positivity. The range for H-score is between 0 and 300. A higher score refers to stronger staining of a particular marker.
Time Frame: Baseline up to 18 Months
Population: Biomarker analysis set: all enrolled participants who had baseline samples submitted as per Institutional Review Board/Independent Ethics Committee approval and participant consent. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measures and "number analyzed" signifies participants evaluable at specific rows.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 13
Score on a scale
  Cytoplasm: AKT: at baseline: number analyzed (Participants) | 11
  Cytoplasm: AKT: at baseline | 99.1 (77.90)
  Cytoplasm: AKT: at Cycle 1 Day 8: number analyzed (Participants) | 10
  Cytoplasm: AKT: at Cycle 1 Day 8 | 123.8 (77.83)
  Cytoplasm: CC3: at baseline: number analyzed (Participants) | 12
  Cytoplasm: CC3: at baseline | 22.1 (28.86)
  Cytoplasm: CC3: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Cytoplasm: CC3: at Cycle 1 Day 8 | 17.9 (27.41)
  Cytoplasm: EGFR: at baseline | 190.4 (113.11)
  Cytoplasm: EGFR: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Cytoplasm: EGFR: at Cycle 1 Day 8 | 184.4 (113.01)
  Cytoplasm: ERK: at baseline | 148.1 (74.26)
  Cytoplasm: ERK: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Cytoplasm: ERK: at Cycle 1 Day 8 | 126.5 (63.80)
  Cytoplasm: HER2: at baseline: number analyzed (Participants) | 11
  Cytoplasm: HER2: at baseline | 36.8 (52.60)
  Cytoplasm: HER2: at Cycle 1 Day 8: number analyzed (Participants) | 10
  Cytoplasm: HER2: at Cycle 1 Day 8 | 43.0 (49.51)
  Cytoplasm: HER3: at baseline | 60.6 (62.49)
  Cytoplasm: HER3: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Cytoplasm: HER3: at Cycle 1 Day 8 | 50.2 (42.41)
  Cytoplasm: pEGFR: at baseline | 101.2 (72.01)
  Cytoplasm: pEGFR: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Cytoplasm: pEGFR: at Cycle 1 Day 8 | 115.6 (56.35)
  Cytoplasm: pEGFR: ratio to baseline: number analyzed (Participants) | 11
  Cytoplasm: pEGFR: ratio to baseline | 1.0 (0.47)
  Cytoplasm: MET: at baseline: number analyzed (Participants) | 12
  Cytoplasm: MET: at baseline | 70.0 (37.31)
  Cytoplasm: MET: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Cytoplasm: MET: at Cycle 1 Day 8 | 81.6 (54.84)
  Cytoplasm: pAKT: at baseline: number analyzed (Participants) | 12
  Cytoplasm: pAKT: at baseline | 41.9 (51.71)
  Cytoplasm: pAKT: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Cytoplasm: pAKT: at Cycle 1 Day 8 | 31.4 (54.78)
  Cytoplasm: pERK: at baseline | 103.3 (46.36)
  Cytoplasm: pERK: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Cytoplasm: pERK: at Cycle 1 Day 8 | 88.3 (41.51)
  Cytoplasm: pHER2: at baseline: number analyzed (Participants) | 11
  Cytoplasm: pHER2: at baseline | 81.6 (31.79)
  Cytoplasm: pHER2: at Cycle 1 Day 8: number analyzed (Participants) | 10
  Cytoplasm: pHER2: at Cycle 1 Day 8 | 78.5 (39.37)
  Cytoplasm: pMET: at baseline: number analyzed (Participants) | 12
  Cytoplasm: pMET: at baseline | 0.0 (0.00)
  Cytoplasm: pMET: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Cytoplasm: pMET: at Cycle 1 Day 8 | 0.0 (0.00)
  Membrane: EGFR: at baseline | 258.3 (60.41)
  Membrane: EGFR: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Membrane: EGFR: at Cycle 1 Day 8 | 209.4 (99.88)
  Membrane: HER2: at baseline: number analyzed (Participants) | 11
  Membrane: HER2: at baseline | 8.2 (24.01)
  Membrane: HER2: at Cycle 1 Day 8: number analyzed (Participants) | 10
  Membrane: HER2: at Cycle 1 Day 8 | 4.3 (8.58)
  Membrane: HER3: at baseline | 12.2 (27.29)
  Membrane: HER3: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Membrane: HER3: at Cycle 1 Day 8 | 9.6 (16.09)
  Membrane: MET: at baseline: number analyzed (Participants) | 12
  Membrane: MET: at baseline | 66.3 (71.26)
  Membrane: MET: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Membrane: MET: at Cycle 1 Day 8 | 53.9 (57.83)
  Membrane: pEGFR: at baseline | 5.8 (14.27)
  Membrane: pEGFR: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Membrane: pEGFR: at Cycle 1 Day 8 | 4.5 (7.27)
  Membrane pHER2: at baseline: number analyzed (Participants) | 11
  Membrane pHER2: at baseline | 1.6 (2.57)
  Membrane pHER2: at Cycle 1 Day 8 | 5.8 (9.28)
  Membrane: pMET: at baseline: number analyzed (Participants) | 12
  Membrane: pMET: at baseline | 0.0 (0.00)
  Membrane: pMET: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Membrane: pMET: at Cycle 1 Day 8 | 0.0 (0.00)
  Nucleus: AKT: at baseline: number analyzed (Participants) | 11
  Nucleus: AKT: at baseline | 87.5 (67.31)
  Nucleus: AKT: at Cycle 1 Day 8: number analyzed (Participants) | 10
  Nucleus: AKT: at Cycle 1 Day 8 | 111.8 (72.93)
  Nucleus: ERK: at baseline | 152.3 (95.93)
  Nucleus: ERK: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Nucleus: ERK: at Cycle 1 Day 8 | 117.5 (73.69)
  Nucleus: pAKT: at baseline: number analyzed (Participants) | 12
  Nucleus: pAKT: at baseline | 40.6 (53.37)
  Nucleus: pAKT: at Cycle 1 Day 8: number analyzed (Participants) | 11
  Nucleus: pAKT: at Cycle 1 Day 8 | 19.1 (38.07)
  Nucleus: pERK: at baseline | 152.7 (88.08)
  Nucleus: pERK: at Cycle 1 Day 8: number analyzed (Participants) | 12
  Nucleus: pERK: at Cycle 1 Day 8 | 144.8 (76.57)

16. Secondary Outcome: H-Score at Ratio to Baseline for Paired Biopsy Biomarkers
Description: as for outcome 15
Time Frame: Baseline up to 18 Months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dacomitinib 45 mg
Number analyzed (Participants) | 13
Ratio
  Cytoplasm: AKT: number analyzed (Participants) | 9
  Cytoplasm: AKT | 2.0 (3.03)
  Cytoplasm: CC3: number analyzed (Participants) | 8
  Cytoplasm: CC3 | 1.0 (0.63)
  Cytoplasm: EGFR: number analyzed (Participants) | 10
  Cytoplasm: EGFR | 1.0 (0.17)
  Cytoplasm: ERK: number analyzed (Participants) | 12
  Cytoplasm: ERK | 0.9 (0.29)
  Cytoplasm: HER2: number analyzed (Participants) | 4
  Cytoplasm: HER2 | 0.7 (0.50)
  Cytoplasm: HER3: number analyzed (Participants) | 11
  Cytoplasm: HER3 | 0.7 (0.60)
  Cytoplasm: pEGFR: number analyzed (Participants) | 11
  Cytoplasm: pEGFR | 1.0 (0.47)
  Cytoplasm: MET: number analyzed (Participants) | 9
  Cytoplasm: MET | 1.2 (0.44)
  Cytoplasm: pAKT: number analyzed (Participants) | 5
  Cytoplasm: pAKT | 0.3 (0.28)
  Cytoplasm: pERK: number analyzed (Participants) | 11
  Cytoplasm: pERK | 0.9 (0.35)
  Cytoplasm: pHER2: number analyzed (Participants) | 9
  Cytoplasm: pHER2 | 0.8 (0.42)
  Membrane: EGFR: number analyzed (Participants) | 12
  Membrane: EGFR | 0.8 (0.33)
  Membrane: HER2: number analyzed (Participants) | 1
  Membrane: HER2 | 0.3 (NA) — Standard deviation could not be calculated due to 1 participant.
  Membrane: HER3: number analyzed (Participants) | 5
  Membrane: HER3 | 0.6 (0.50)
  Membrane: MET: number analyzed (Participants) | 8
  Membrane: MET | 0.8 (0.41)
  Membrane: pEGFR: number analyzed (Participants) | 4
  Membrane: pEGFR | 2.5 (4.33)
  Membrane pHER2: number analyzed (Participants) | 4
  Membrane pHER2 | 4.3 (4.50)
  Nucleus: AKT: number analyzed (Participants) | 8
  Nucleus: AKT | 2.8 (4.73)
  Nucleus: ERK: number analyzed (Participants) | 10
  Nucleus: ERK | 1.1 (1.38)
  Nucleus: pAKT: number analyzed (Participants) | 7
  Nucleus: pAKT | 0.3 (0.59)
  Nucleus: pERK: number analyzed (Participants) | 10
  Nucleus: pERK | 0.9 (0.33)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Dacomitinib 45 mg
Serious Adverse Events (participants affected / at risk) | 20/69
Other Adverse Events (participants affected / at risk) | 68/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib 45 mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Disease progression (General disorders) | 4
Brain abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib 45 mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Blepharitis (Eye disorders) | 3
Conjunctival irritation (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 6
Dry eye (Eye disorders) | 2
Entropion (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye oedema (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 2
Eyelids pruritus (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Vision blurred (Eye disorders) | 3
Visual impairment (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Aptyalism (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 58
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 8
Eructation (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 3
Lip dry (Gastrointestinal disorders) | 2
Lip haemorrhage (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Odynophagia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Saliva altered (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 10
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 5
Chills (General disorders) | 4
Face oedema (General disorders) | 3
Fatigue (General disorders) | 35
Influenza like illness (General disorders) | 1
Irritability (General disorders) | 1
Local swelling (General disorders) | 1
Mucosal inflammation (General disorders) | 11
Oedema peripheral (General disorders) | 6
Performance status decreased (General disorders) | 1
Pyrexia (General disorders) | 5
Candidiasis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Groin infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 12
Pneumonia (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 6
Skin infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 2
Eye penetration (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
Weight decreased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 3
Motor dysfunction (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
VIIth nerve paralysis (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 7
Libido decreased (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 52
Dry skin (Skin and subcutaneous tissue disorders) | 34
Erythema (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Exfoliative rash (Skin and subcutaneous tissue disorders) | 17
Granuloma skin (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 6
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 11
Rash erythematous (Skin and subcutaneous tissue disorders) | 5
Scab (Skin and subcutaneous tissue disorders) | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Intra-abdominal haematoma (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.